CLINICAL TRIAL: NCT06846957
Title: ESSENCE Study: E-health Self Symptom AssEssmeNt As a Front Door and Facilitator of CarE, Portugal
Brief Title: ESSENCE is a Quality Improvement Study That Evaluates the Impact of Ada's AI-powered Core Symptom Assessment Technology on Clinical Workflow and Individual Healthcare Guidance, Following the November 2021 Integration of the Tool Into the CUF Hospital Network. Study Duration Nov 2024-Oct 2025
Acronym: ESSENCE
Status: Completed | Type: Observational
Sponsor: Ada Health GmbH (Industry)
Collaborators: Academia Cuf Descobertas (Network); Hospital CUF Descobertas, Lisbon, Portugal (Unknown); CUF Tejo Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: EudraCT number: 2022-000067-42
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Symptom Assessment
Keywords: digital health; AI; patient outcomes; symptom assessment application; symptom checker; Ada; CUF; Portugal; ESSENCE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A 1.5.1 Study title ESSENCE Study: E-health Self Symptom assEssmeNt as a front door and facilitator of CarE

A 1.5.2 Investigational device 'Ada Assess' (CE-marked), 'Ada Connect' (a software integrating with CE-marked medical devices), and 'Ada Handover' (a CE-marked component of the 'Ada Assess' product that shares the same version number).

A 1.5.3 The Ada Health-CUF Integration To improve MyCUF service, CUF partnered with Ada Health, a symptom assessment application in which the patient can enter their/their children's symptoms, answer follow-up questions, and receive a list of potential causes, additional health information, and advice on if, when, and where to seek medical care.

A 1.5.4 Study design ESSENCE is a Quality Improvement (QI) study that evaluates the impact of Ada's AI-powered core symptom assessment technology on clinical workflow and individual healthcare guidance, following the November 2021 integration of the tool into the CUF hospital network.

A 1.5.5 Study objectives

The study has 3 main objectives:

1. Assess the clinician-perceived appropriateness of the Ada symptom assessment report.
2. Examine the impact of the Ada symptom assessment report on consultation efficiency.
3. Evaluate the effect of the Ada symptom assessment on patients' health-seeking behavior.

A 1.5.6 Primary and secondary endpoints

The primary endpoints of the study include:

(i) Appropriateness of the urgency advice provided by Ada and (ii) appropriateness of the Ada symptom assessment report, including factors such as reasonability of suggested conditions, completeness of symptom/medical history, agreement of medical problem summarized in the report with patient-HCP consultations, and the proportion of condition suggestions matching the main diagnosis.

Secondary endpoints encompass:

(i) The impact of the Ada Symptom Assessment Report on consultation efficiency, including changes in consultation activity distribution and resulting time saved for specific activities, (ii) the influence of the Ada assessment on patients' health-seeking behavior, including changes in health-seeking intent and behavior before and after checking their symptoms, (iII) assessment of the impact of the Ada assessment on the psychological well-being of patients, (iv) an exploration of health economic benefits resulting from the use of Ada's symptom assessment, and (v) an exploration of addition of large language models (LLMs) to the SC to: measure improvements in diagnostic accuracy measure improvements in the quality of differential diagnosis list measure improvements in safety and appropriateness of urgency advice These endpoints collectively aim to provide comprehensive insights into the impact and effectiveness of Ada's symptom assessment tool within the healthcare system.

A 1.5.7 Study size & duration Over the estimated 12 -month study period from November 2023 to October 2024, the study aims to enrol 143 CUF patients as study subjects, who consent both to 'Ada Handover' and to study participation and schedule a consultation with a CUF physician. The study subject number calculation determined that 143 subjects are required to enable primary endpoint analysis, and the study shall continue until this number of subjects for primary endpoint analysis are recruited. It is anticipated that not all patients consenting to participate in the study will schedule an appointment with a CUF physician and therefore no primary endpoint analysis can be performed. For these patients, only the routinely collected information of the symptom assessment flow will be stored in the dedicated electronic data capturing system and used for secondary endpoint/additional data analysis. We will also gather health-seeking behavior of these patients via a follow-up email which will be used for secondary endpoint analyses. It is also anticipated that some participating physicians may miss patients eligible for the primary endpoint due to technical or other difficulties. In this event, only relevant data points will be collected at the end of the study.It is estimated that around 2000 patients will be enrolled to ensure 143 patients are eligible for primary endpoint analysis.

If it is not possible to recruit the target subject number in 12 months, the PI and Sponsor will discuss whether the study shall terminate before this target is reached, and this will be discussed with the Ethics Committee if required. If the target patient recruitment number is reached earlier than the estimated 12 -month study period, the sponsor and Principal Investigator (PI) will discuss increasing the number of enrolled patients to provide additional power for potential sub-analyses. No data will be analysed for those CUF users who did not consent to 'Ada Handover' or study participation.

DETAILED DESCRIPTION:
A 1.5.4 Study design ESSENCE is a Quality Improvement (QI) study that evaluates the impact of Ada's AI-powered core symptom assessment technology on clinical workflow and individual healthcare guidance, following the November 2021 integration of the tool into the CUF hospital network.

A 1.5.5 Study objectives

The study has 3 main objectives:

Assess the clinician-perceived appropriateness of the Ada symptom assessment report.

Examine the impact of the Ada symptom assessment report on consultation efficiency.

Evaluate the effect of the Ada symptom assessment on patients' health-seeking behavior.

A 1.5.6 Primary and secondary endpoints

The primary endpoints of the study include:

(i) Appropriateness of the urgency advice provided by Ada and (ii) appropriateness of the Ada symptom assessment report, including factors such as reasonability of suggested conditions, completeness of symptom/medical history, agreement of medical problem summarised in the report with patient-HCP consultations, and the proportion of condition suggestions matching the main diagnosis.

Secondary endpoints encompass:

(i) The impact of the Ada Symptom Assessment Report on consultation efficiency, including changes in consultation activity distribution and resulting time saved for specific activities, (ii) the influence of the Ada assessment on patients' health-seeking behaviour, including changes in health-seeking intent and behaviour before and after checking their symptoms, (iII) assessment of the impact of the Ada assessment on the psychological well-being of patients, (iv) an exploration of health economic benefits resulting from the use of Ada's symptom assessment, (v) an exploration of addition of large language models (LLMs) to the SC to: measure improvements in diagnostic accuracy measure improvements in the quality of differential diagnosis list measure improvements in safety and appropriateness of urgency advice These endpoints collectively aim to provide comprehensive insights into the impact and effectiveness of Ada's symptom assessment tool within the healthcare system.

A 1.5.7 Study size & duration Over the estimated 12 -month study period from November 2023 to October 2024, the study aims to enrol 143 CUF patients as study subjects, who consent both to 'Ada Handover' and to study participation and schedule a consultation with a CUF physician. The study subject number calculation determined that 143 subjects are required to enable primary endpoint analysis, and the study shall continue until this number of subjects for primary endpoint analysis are recruited. It is anticipated that not all patients consenting to participate in the study will schedule an appointment with a CUF physician and therefore no primary endpoint analysis can be performed. For these patients, only the routinely collected information of the symptom assessment flow will be stored in the dedicated electronic data capturing system and used for secondary endpoint/additional data analysis. We will also gather health-seeking behaviour of these patients via a follow-up email which will be used for secondary endpoint analyses. It is also anticipated that some participating physicians may miss patients eligible for the primary endpoint due to technical or other difficulties. In this event, only relevant data points will be collected at the end of the study. It is estimated that around 2000 patients will be enrolled to ensure 143 patients are eligible for primary endpoint analysis.

If it is not possible to recruit the target subject number in 12 months, the PI and Sponsor will discuss whether the study shall terminate before this target is reached, and this will be discussed with the Ethics Committee if required. If the target patient recruitment number is reached earlier than the estimated 12 -month study period, the sponsor and Principal Investigator (PI) will discuss increasing the number of enrolled patients to provide additional power for potential sub-analyses. No data will be analysed for those CUF users who did not consent to 'Ada Handover' or study participation.

A.2 Identification and description of the investigational device This is a Post-Market study conducted under a Quality Improvement framework for 'Ada Assess,' 'Ada Connect' and 'Ada Handover', as integrated with the myCUF app. The relevant software has all required regulatory approval and is CE-marked and will already be integrated with the myCUF app and used by patients before the commencement of the clinical study.

A2.1 Manufacturer details Name: Ada Health GmbH Address: Neue Grünstrasse 17 10179 Berlin, Germany

Phone: +49 30 403 67 390 Website: www.ada.com Email: hello@ada.com A 2.2 General Description Name of the device: 'Ada Assess' (CE-marked), 'Ada Connect' (a software integrating with CE-marked medical devices), and 'Ada Handover' (a CE-marked component of the 'Ada Assess' product that shares the same revision number) and medical device accessory to Ada Assess: SDK.

The software version numbers used in the Clinical Investigation will be recorded in the Trial Master File.

'Ada Assess' is a Class IIa CE-marked medical device software application. 'Ada Assess' runs as an embedded iFrame or modal window application that is integrated into the clients' website or mobile application. It is accessible from both desktop and mobile devices. It supports all browser types and is independent of operating systems. Ada Assess requires an active internet connection as it does not function offline. That allows users to obtain relevant information about possible causes of their health symptoms by using medical intelligence and probabilistic reasoning. It was embedded in both mobile and web applications of CUF using software development kits (SDKs). By initiating an assessment, the user is requested to enter relevant information about themselves. Some of their relevant information can be directly accessed from CUF and their Electronic Health Record (EHR) via Single Sign-On (SSO). Following this, they are guided through a logical sequence of questions, intended to identify possible medical conditions that cause the specified symptoms or health findings. At the end of the assessment the user is provided with a report, referred to as an "assessment report", that lists probable causes behind their symptoms and explains actionable next steps as well as care navigation options from the CUF network. The assessment report can be downloaded as a PDF document. The user can also choose to share their assessment report with a doctor or CUF.

A 2.3. Use Specification A 2.3.1 Intended Use "Ada Assess is a personal health assessment application designed for providing personal health insights and information. The application is intended to enable users to enter symptoms and other relevant health information or to access relevant health information from the user's health record or health provider and, through the use of medical intelligence and probabilistic reasoning, to identify possible causes for health findings and symptoms. It also provides information about possible causes and next steps and can allow the user to share this information with their doctor or healthcare provider (for informing the doctor/health care provider, not to drive diagnostic decision making by the doctor/health care provider).

Note: Ada Assess is not a substitute for advice from a healthcare professional. Should the symptoms persist, get worse or if additional symptoms are noticed, then it is recommended that the user immediately seeks professional medical attention." A2.3.2 Indications for use Ada Assess does not have any further specific indication for use. Ada Assess can consider thousands of symptoms and health findings and includes a library with thousands of conditions.

A 2.3.3 Intended Users The application is designed for use by individuals over the age of 16. Individuals over the age of 16 may carry out health assessments for others (e.g. family members) including children, provided they are the child's legal guardian (the user must agree to this in the Terms and Conditions of the application).

General Training requirements No special training is required to use 'Ada Assess' to carry out a symptom assessment by patients/users.

Note: Training will be provided to all relevant physicians and other staff on roll-out of the system to the healthcare system. Additionally, investigation-specific training will be provided to all relevant health care practitioners, so that they are familiar with 'Ada Assess', 'Ada Connect' and 'Ada Handover', the clinical investigation protocol, and the eCRFs.

A 2.3.4 Contraindications 'Ada Assess' must not be used under critical and emergency situations. A 2.3.5 Location and Conditions for Use 'Ada Assess' runs as an embedded iFrame or modal window application that is integrated into CUFs website or the myCUF mobile application. It is accessible from both desktop and mobile devices. It supports all browser types and is independent of operating systems. Ada Assess requires an active internet connection as it does not function offline.

A2.4 Operating principles and functions A2.4.1 Key functions The key function of Ada Assess is the intelligent health findings assessment, with further information provided as part of the assessment report, such as the actionable next steps and general description of the conditions.

Upon users' first access to the Ada Assess app, the app elicits some basic personal information from them (name, date of birth, gender) and some basic risk factors (Diabetes, Hypertension, smoking status, pregnancy). The app may also ask for some additional general health information or inquire about the intent of doing a health assessment. After the user has answered all questions, the Ada Assess application begins the assessment by asking the user to state any current symptoms and other health findings. It qualifies the information collected by asking for and establishing attributes such as acuity and time since onset. Ada Assess then asks the user about the presence or absence of a series of medical findings related to the presented symptoms, using custom probabilistic reasoning technology. This technology reviews multiple pieces of data provided by the user to output probabilities. This way it can consider a variety of conditions and diseases to make a health assessment, using the question flow to rule out some causes and pursue other possible causes, finishing by providing the user a report with a list of the most likely conditions that are causing their findings.

This assessment report can be downloaded by the user as a PDF file. Ada Assess also contains an optional 'Handover' feature that can share this report with the user's doctor or CUF as their healthcare provider.

The shared report aims to inform the patient's doctor/healthcare provider of the information the patient has received from 'Ada Assess'. This report includes the information shown to the patient after completing the symptom assessment and the questions the user was asked by Ada Assess, including their self-reported complaints and suggested conditions that may be causing these symptoms. It is not intended to drive diagnostic decision-making or to dictate or override the diagnostic workup planned by the treating physician. Ada Assess uses Brazilian Portuguese for the question flow and the assessment report.

A 2.4.2 Additional interactions and interfaces A 2.4.2.1 Connect 'Ada Assess' is integrated with an additional software unit from Ada Health's system, known as Connect. Connect is not part of the medical device and is technically and by design a separate unit from the Ada Assess medical device.

After completion of a health assessment in Ada Assess and the delivery of an assessment report, Connect provides the user an opportunity to review and select relevant partner healthcare services, studies or information. Connect is intended to inform laypersons around the possible options for CUFs healthcare services based on the advice level and possible causes. Care options are visible after the user completes a health assessment; next to the possible causes. These options can then be filtered by location, relevance and more. Currently, the options Call Ambulance, Emergency Care or Telemedicine Consultation with a General Practitioner or Paediatrician will be shown to the user.

A 2.4.2.2 Single Sign-On via the Smart Auth service 'Ada Assess' was also integrated with an additional software unit from Ada Health's system, known as Smart Auth. Smart Auth is not part of the medical device and is technically and by design a separate unit from the Ada Assess medical device.

As mentioned above, the application requires some basic personal and risk factor information in order to provide the health assessment. CUF as the healthcare provider was able to choose to provide some of this demographic and risk factor information automatically via single sign-on (SSO) using the Smart Auth service.

A 2.4.2.3 FHIR interoperability The assessment report produced by 'Ada Assess' will also be converted into the Fast Healthcare Interoperability Resources (FHIR) format to allow compatibility with partner systems and electronic health records (EHR) when sent via the Handover feature. FHIR interoperability is used for general interfacing of the medical device and non-medical device aspects of Ada Health's system and the partner system, and as functionality for general secure information transfer, this interoperability is not classified within the 'Ada Assess' medical device.

A 2.4.3 Safety-related features All assessments provided by 'Ada Assess' include a clear statement that the results do not constitute an official medical diagnosis and that the user is advised to seek professional help if they are seriously concerned about their symptoms or health findings.

A 3 Justification for the design of the clinical investigation A 3.1 An evaluation of the results of the relevant pre-clinical testing/assessment and prior clinical investigations This medical device software to be evaluated in this clinical investigation has been on the market as a CE marked Class IIa medical device and has a valid CE-mark.

Externally validated and safety demonstrated: Ada Health's assessment technology has been clinically validated through numerous scientific studies to be accurate, safe, and convenient to use by medically untrained people. See https://ada.com/studies/ for a detailed list of published peer-reviewed studies.6-12 A UK study with different digital assessment applications and general practitioners (GPs) found Ada Health's assessment technology to be the most accurate and safe digital tool across 200 clinical vignettes representing a broad spectrum of medical conditions and within the range of GPs.6 In the same study, a safety rate of the app's urgency advice was 97% which lay within 1 SD of the compared GPs.6 A study using Ada Health's assessment technology adapted for use by medical professionals found the assessment to be 94.7% safe in patients presenting to the Emergency Department in Marburg, Germany.12 In another Emergency Department study, Handover of the Ada Symptom Assessment Report was evaluated with 75% of patients, 73% physicians and 100% nurses considering the tool useful in facilitating conversation and for some medical specialism time-saving.13 The clinical benefit through efficiency saving potential of HCP-handover of the symptom and history information in the assessment report was also demonstrated in a simulation study.14 Ada Health's symptom assessment is quick to complete for users, 3.6 minutes on average. Studies found the assessment was highly usable7 and highly accepted by patients.8 In addition to peer-reviewed external validation studies, Ada Health is internally generating pre-clinical data based on several hundred test cases which were created by medical professionals blinded to the work of Medical Knowledge and Medical Intelligence teams to test the accuracy of the condition suggestions and advice level suggestions. These tests are being carried out before every release (i.e. with every change to 'Ada Assess' and/or the shared software algorithm platform, the 'Ada Medical Intelligence') and on a continuous basis throughout the lifetime of the device. The predefined acceptance level of condition and urgency advice have to be met to pass these tests.

A.4 Benefits and risks of the investigational device, clinical procedure, and clinical investigation A4.1 Anticipated clinical benefits. Intended Benefit - Timely and accurate symptom assessment for the lay user: 'Ada Assess' provides the lay-user/patient an initial assessment of their symptoms and provides a list of possible conditions (condition-suggestions) and guidance to appropriate next steps in engagement with HCPs (e.g., an indication of how soon they should see their GP, to support decision-making). This function is similar to the assistance a patient traditionally obtained by reference to a family medical encyclopaedia and is similar to the assistance patients often now obtain through an internet search engine of symptoms; the advantage is the self-tailored curated medical-reasoning-based information and highly usable interface.

Intended Benefit - User's peace of mind: The ability to have personalised, immediate, mobile, personalised health information (in non-emergency situations) 24/7 potentially provides peace of mind.

Intended Benefit - Health awareness: Personal symptom assessment, complemented with identification of appropriate next steps (including medical support), helps patients to take ownership of their health (both physical and mental) by providing better health insights and information. This has motivational effects leading to more self-management and care and increased health awareness.

Intended Benefit - Health information access: Free access to reliable healthcare information is of fundamental importance and benefit.

Intended Benefit - Less common and rare disease identification: We have evidence that for less-common and rare disease patients, the 'Ada Health Assessment' has the potential to assist users in arriving at a timely HCP medical diagnosis. Less common and rare disease diagnoses remain a challenge for patients, doctors, and healthcare systems and are often delayed by years. On average, rare disease patients wait for about 6 years from the onset of symptoms to an accurate diagnosis while in the process of going through a diagnostic odyssey10. Lack of scientific knowledge and quality information on the disease may lead to misdiagnosis, a part of the challenge in identifying patients with rare diseases. The 'Ada Medical Intelligence' has shown potential for making patients aware of these uncommon and rare conditions and thus supporting individuals' communication and engagement with HCPs, with the potential for assistance in arriving at a timely diagnosis. This not only has the potential to improve the quality of life for these patients but also has the potential to reduce unnecessary consultations and in turn reduce the substantial costs for both the patients and healthcare systems.10 Note: the prototype clinical decision support system 'Ada DX DDSS Prototype Application' assessed in (Ronicke et al., 2019) has a different Intended Purpose than the 'Ada Assess', but it is a 'similar device' using the same underlying 'Ada Medical Intelligence' as 'Ada Assess'.

Intended Benefit - Potential to engage the patient in the diagnostic journey with the HCP: Correct and timely diagnosis plays a very important role in disease identification and its management. The traditional view has often been that diagnosis is a one-sided process delivered to the patient with their role in the process ending at describing their symptoms and family history. In reality and increasingly, the patient is involved in their journey to a diagnosis. Patients' access to quality information about their symptoms and predisposing factors is essential. 'Ada Assess' provides this information. User/patient feedback evidence shows that, in the view of the patient and of HCPs, that the 'Ada Health Assessment Report' can assist in pre-assessment of patients by gathering relevant history and comprehensive information about presenting symptoms.

Intended Benefit - Potential for appointment prioritisation: Pre-assessment of patients (based on their presenting symptoms) can help clinicians/practices to better identify the need for intervention and can help prioritise patient appointments.

Intended Benefit - Facilitation of interaction between the user and their health care professional: 'Ada Assess' supports the user/patient to perform an initial self-assessment of their symptoms and provides a highly usable easily interpretable symptom-level health assessment. This report can, if the patient wishes, be shared with the HCP and can facilitate communication - speeding communication of symptom information, freeing up time for quality communication between the HCP and patient) and/or increasing health care provision efficiency. Sharing can be facilitated via paper or electronic means (PDF or via making the report available to the HCP via secure FHIR connection to the patient's Electronic Medical Record, with the manner of display of the information designed and controlled by the healthcare provider systems designers and administrators).

Potential Benefit - Cost-benefit: 'Ada Assess' helps individuals identify and understand the possible cause of their symptoms and supports them in identifying appropriate next steps including medical support. In non-emergency situations, this can lead to a reduction in the number of visits to primary health care providers, thus having a positive financial impact.

Potential Benefit - Reduced waiting room time (and associated stress): For some simple minor and non-emergency situations provided information can help the patient decision making to seek an appropriate alternative to immediate HCP visit - e.g. where a pharmacy visit is more appropriate. This has the potential to reduce the stress associated with obtaining a GP appointment and reduce the stress (and potential for nosocomial infection) associated with unnecessary time spent in the GP's practice waiting and consultation rooms. This has also potential to free up HCP resources for other patients and reduce HCP and Payer costs.

A4.2 Anticipated adverse device effects Use of digital health tools may be related to increased health anxiety, particularly if the conditions suggested to the user include distressing or sensitive conditions Use of digital health tools may be related to increased self-surveillance and the normalisation of health-seeking behaviour.

Use of the application could potentially increase the time to seek medical care to finish the assessment which could be a risk to patients' health in case of emergency. It is stated that the product should not be used in case of an obvious emergency and has been designed to stop the assessment if clear emergency symptoms were entered.

It is possible that the provided urgency advice is lower than considered appropriate by clinicians.

It is possible that for healthcare professionals (HCPs) reviewing the Handover report, the information received could conflict with their own clinical perspective on the patient's medical problem, and therefore result in either a challenging situation to explain to the patient (with respect to the different information provided on the medical problem).

iIf the Handover report is not as medically accurate as anticipated, or if system technical difficulties occur too frequently , this could lead to a loss of HCP confidence in the system.

A4.3 Risks associated with participation in the clinical investigation A4.3.1 Study type: interventional / non-interventional

An important note on the study type:

This clinical investigation has no intervention for patients. There is no change made to patients' standard of care for those patients who consent to study participation. There are no consequences for patients who decide not to participate or who initially consent to participate and then later withdraw their content. 'Ada Assess' is a Class IIa medical device already in use prior to the clinical investigation; it continues to be used in its normal intended purpose with no additional procedures for patients, and therefore, no burdensome additional procedures for patients, given they consent to participate. We may reach out to individual patients who did not book a consultation with CUF after using Ada or if we have specific enquiries about their healthcare journey. However, there is no obligation to respond to this message.

Physicians who consent to participate in the study (via a full clinical studies informed consent process) only experience two minor changes to their normal working practices; neither of these changes are burdensome, as they relate to the completion of simple eCRF questionnaires:

The consenting physicians complete one simple baseline eCRF questionnaire after they consent to participate in the study.

The consenting physicians complete another simple eCRF questionnaire for each consenting patient either (i) after the consultation with that patient or (ii) at the end of the working day or (iii) retrospectively at the end of the study period for missed patients for relevant data points.

This questionnaire asks about the performance and value of the 'Ada Assess' system. All consenting physicians will be fully trained in the clinical investigation and in the eCRFs prior to study initiation.

As this is therefore, with respect to patients, an observational post-market clinical investigation (exploring the medical device in its normal intended use, with consent, and with no additional procedures, burdensome or otherwise) conducted as a Quality Improvement data-gathering activity. The usual patient journey is monitored without any study-related changes. We have examined the entire CUF patient journey, and we have been unable to identify any additional risk for patients who participate in this clinical investigation. In case the patient decides to use the myCUF App and the symptom assessment application, they could potentially (but are highly unlikely to) experience some of the anticipated adverse device effects listed above, but this will not be due to an intervention associated with the clinical investigation, as this system is part of normal care for any patient that chooses to use it. There is no intervention with respect to consenting participating patients in this clinical investigation, and any adverse effects that could occur are related to the usual product use in regard to the probability of occurrence or the severity.

Ada Health had an email consultation with INFARMED on 27-28 December 2021. We understand that INFARMED considers the overall investigation to be interventional because consenting participating physicians will complete two simple eCRF questionnaires. We understand that because this is the local legal definition of interventional, the overall study classification must be considered 'interventional', and the documentation requirements of interventional MDR studies must be fulfilled.

Nonetheless, the risk assessment of the study is as follows:

Patient involvement: this aspect of the study is observational/interventional with respect to patient involvement with no clinical risk associated with the clinical investigation [The overall clinical investigation is defined as interventional, as consenting participating physicians complete two simple eCRF questionnaires; however, there are no burdensome additional procedures for consenting participating patients (see Section 4.3.1)]. The participating patients consent to clinical data sharing within the study; this includes an identified hazard of the inadvertent sharing of this data if clinical investigation data protections systems were to fail. A validated Electronic Data Capture (EDC) system will be used; all EDC procedures follow GDPR requirements for patient consent and have been designed to minimise the risk of inadvertent data loss/release. After the implementation of all mitigation measures as described above, the risk of a data security compromise is extremely unlikely.

There are no other identified risks with respect to patient participation. Physician involvement: No risks have been identified associated with the physician completion of either of the clinical investigation eCRFs.

A4.4 Steps that will be taken to control or mitigate the risks. If the patient presents with suicidal ideation, hemiparesis, haematemesis, or other serious symptoms during the Question Flow, the assessment will immediately stop and inform the user that this is a serious condition and they need to seek medical attention right away. The user can still proceed with the assessment if they choose to. Note: this is not a specific clinical investigation associated risk; it is, instead, a general risk associated with the use of the 'Ada Assess' medical device, which is already in routine use, for patients who choose to use it, within the CUF healthcare system.

A4.5 Rationale for benefit-risk ratio. This study's purpose is monitoring, evaluation and quality improvement of a system already placed on the market and already risk assessed as having an acceptable benefit/risk profile for the market. As participation in this clinical investigation poses no additional risks, we consider the burden/risks of this study very low.

A5. Objectives and hypothesis of the clinical investigation A 5.1 The purpose of the clinical investigation, claims for clinical performance, effectiveness or safety of the investigational device to be verified.

Using a Quality Improvement (QI) framework, this study will monitor the real-world performance of the Ada Health-CUF integration with a focus on clinician-perceived appropriateness and the impact of the Ada symptom assessment report on consultation efficiency and the effect on patients' health-seeking behavior.

Regarding its defined intended purpose the product has been implemented to provide patients with information on their symptoms with possible conditions causing them and about possible next steps (e.g. assistance of patients in choosing the best healthcare unit for their medical need). This information will be collected in an assessment report which will be available for the patient to download as PDF and to share with their HCP if they wish. The HCP can therefore use the collected information for their medical consultation. All users of the symptom assessment application are routinely being asked one question before and after the assessment. For users consenting to participating in the study, this information will together with the information from the assessment report transferred to the EDC system.

The purpose of this clinical investigation is to evaluate the quality, value, benefit, safety and performance of 'Ada Assess', 'Ada Connect' and 'Ada Handover' for patients and the health care system through positive impact on patient management. The worth of the product is ultimately linked to medical appropriateness and safety of medical information included in the assessment report which will be measured in this clinical investigation. All information collected will be used to identify strengths and weaknesses of the product on which base product changes can be discussed

ELIGIBILITY:
Inclusion Criteria:

* Any individual who is 18 years old or above and utilises the CUF application to evaluate their own symptoms using 'Ada Assess' and who consents to participate in this clinical investigation and to Ada 'Handover'.

Exclusion Criteria:

* Users under the age of 18 years will be excluded. Users who conduct a symptom assessment on behalf of others will be excluded. Users who do not consent to sharing the symptom assessment report with CUF will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual who is 18 years old or above and utilises the CUF application to evaluate their own symptoms using 'Ada Assess' and who consents to participate in this clinical investigation and to Ada 'Handover'.
Sampling Method: Non-Probability Sample
Enrollment: 1470 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of ada's condition report and triage classification | 12 months
  1. Appropriateness of Ada's urgency advice
  2. Appropriateness of the 'Ada Symptom Assessment Report,' considering all information points provided. This will be a composite of ratings on
     1. Reasonability of the suggested conditions,
     2. Completeness rating on symptom/medical history,
     3. Agreement of the medical problem presented in the Assessment Report with the presentation in the patient-HCP consultation

SECONDARY OUTCOMES:
Impact of Ada on patient and physician healthcare behaviours | 12 months
  Impact of the Ada Symptom Assessment Report on consultation efficiency. This will be a composite of ratings on Facilitation of the clinical conversation by the Ada Symptom Assessment Report, Time-saving utility of the Ada Symptom Assessment Report , Usefulness of conditions for the diagnostic workup. Proportion of condition suggestions provided by the Ada Symptom Assessment matching the main diagnosis/discharge diagnosis determined by the treating physician Impact of the Ada Assessment Report on patient's health seeking behaviour measured by comparing intent of patients pre- and post-assessment Psychological impact on patients health as a result of the information provided in the Ada Symptom Assessment determined by the treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Flores, MD, Principal Investigator — CUF hospital Network
Locations (1):
- CUF Hospital Network, Lisbon, Carnaxide, Portugal

IPD SHARING:
Plan to Share IPD: No